CLINICAL TRIAL: NCT00009893
Title: Phase II Trial Of Gemcitabine, 5-Fluorouracil, And Leucovorin In Patients With Measurable Unresectable Or Metastatic Biliary Tract Carcinoma (Intrahepatic, Extrahepatic, Ampulla Of Vater) And Gallbladder Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Unresectable or Metastatic Biliary Tract or Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0042; NCI-2012-02370 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068421 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-02-02; First posted 2004-01-01 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Fluorouracil; Gemcitabine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + leucovorin + fluorouracil (Experimental): Patients receive gemcitabine IV over 30 minutes followed by leucovorin calcium IV and fluorouracil IV over 5-10 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have unresectable or metastatic biliary tract or gallbladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the 6-month survival and overall survival of patients with unresectable or metastatic biliary tract carcinoma or gallbladder cancer treated with gemcitabine, fluorouracil, and leucovorin calcium. II. Determine the tumor response in these patients treated with this regimen. III. Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes followed by leucovorin calcium IV and fluorouracil IV over 5-10 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable or metastatic biliary tract carcinoma (extrahepatic, intrahepatic, or ampulla of Vater) or gallbladder carcinoma Not amenable to combined chemotherapy and radiotherapy CNS metastases that are locally treatable (i.e., lesions treatable with surgery or radiotherapy) allowed if no evidence of progression for at least 4 weeks after completion of treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 3.0 times upper limit of normal (ULN) AST no greater than 5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic or immunologic therapy No prior biologic or immunologic therapy for metastatic disease No concurrent immunotherapy No colony stimulating factors administered concurrently with first course of study therapy, or within 24 hours prior to subsequent courses Chemotherapy: See Disease Characteristics No prior gemcitabine No prior chemotherapy for metastatic disease At least 6 months since prior chemotherapy used as radiosensitization either in the adjuvant setting or for locally advanced disease No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to more than 25% of bone marrow No concurrent radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
survival at 6 months | at 6 months

SECONDARY OUTCOMES:
overall survival | Up to 5 years
tumor response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Alberts SR, Al-Khatib H, Mahoney MR, Burgart L, Cera PJ, Flynn PJ, Finch TR, Levitt R, Windschitl HE, Knost JA, Tschetter LK. Gemcitabine, 5-fluorouracil, and leucovorin in advanced biliary tract and gallbladder carcinoma: a North Central Cancer Treatment Group phase II trial. Cancer. 2005 Jan 1;103(1):111-8. doi: 10.1002/cncr.20753. PMID 15558814